CLINICAL TRIAL: NCT06440044
Title: Recurrence and Bleeding in Colorectal Cancer Patients With Cancer-associated Venous Thrombembolism
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024ZSLYEC-226
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-05

CONDITIONS: Thrombosis, Venous; Colo-rectal Cancer; Bleeding
Keywords: Venous Thrombembolism；Colorectal Cancer；Bleeding
MeSH Terms: conditions — Venous Thrombosis; Colonic Neoplasms; Hemorrhage | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with adverse anticoagulant outcomes: Patients with adverse anticoagulant outcomes in the study period. Adverse anticoagulant outcomes include venous thromboembolism recurrence, major bleeding, and clinical relevant non major bleeding.
  Interventions: Other: Data collection
- Patients without any adverse anticoagulant outcomes: Patients without any adverse anticoagulant outcomes in the study period.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — A prospectively maintained database query of all patients with CRC and VTE was initially performed, and then each patient's electronic record was reviewed for inclusion criteria.

SUMMARY:
Patients with colorectal cancer (CRC) have a higher risk of both venous thromboembolism (VTE) and major bleeding (MB). Patients with CRC are underrepresented in the major trials examining treatment of cancer-associated VTE with anticoagulant.

DETAILED DESCRIPTION:
Patients with colorectal cancer (CRC) have a higher risk of both venous thromboembolism (VTE) and major bleeding (MB). Specifically, a subsequent analysis of the Hokusai study showed that the excess in MB was confined to patients with gastrointestinal cancer. In the RIETE registry, patients with gastrointestinal or genitourinary cancers experienced more bleeding outcomes while patients with brain or lung cancer experienced more thrombotic outcomes. However, in a subgroup analysis of the Caravaggio trial, major gastrointestinal bleeding in patients with CRC was low and similar in both apixaban and LMWH groups. Patients with CRC are underrepresented in the major trials examining treatment of CAT with anticoagulant. Despite concerns that DOACs pose a significant bleeding risk in CRC patients, many patients with CRC are treated with apixaban or rivaroxaban in clinical practice. Balancing risks of thrombosis recurrence and bleeding can be challenging and requires a nuanced, individualized approach to decision making to improve prognosis in this population. The aim of this study is to identify risk factors for recurrence and bleeding in CRC patients with VTE. Deaths, regardless of the mechanism, will also be included in the one year all-cause mortality outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed CRC and symptomatic or incidental VTE who received anticoagulant treatment.
2. CRC patients with VTE treated with an anticoagulant (rivaroxaban or LMWH) for at least six months.

Exclusion Criteria:

1. Participation in this study required active anticoagulant treatment. Apart from this, there were no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed CRC and symptomatic or incidental VTE who received anticoagulant treatment at The Sixth Affiliated Hospital, Sun Yat-sen University from January 2019 to January 2023. VTE was considered cancer-related if the patient had a diagnosis of CRC within six months before or after the VTE diagnosis, any cancer treatment within the previous six months, or recurrent/metastatic cancer regardless of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
recurrent VTE including deep vein thrombosis (DVT) and pulmonary embolism (PE) | From the date of index VTE to VTE recurrence, assessed up to 12 months
  Recurrent DVT had to be confirmed by duplex ultrasonography, venography, CT, or MRI. Recurrent PE was confirmed by CT, MRI, conventional pulmonary angiography, or VQ (ventilation/perfusion) imaging. Fatal PE had to be based on objective diagnostic testing, autopsy, or death that could not be attributed to a documented cause and for which PE/DVT could not be ruled out (unexplained death). Incidental VTE recurrence had to be identified via surveillance-related imaging. To be classified as a recurrent event, a new filling defect had to be evident on the second study, not appreciated on the original images, or an interval study clearly showing thrombus resolution.
Major Bleeding (MB) | From the date of index VTE to MB occurrence, assessed up to 12 months
  MB was defined as overt bleeding plus a hemoglobin decrease of ≥ 2 g/dL after the incident, requirement for transfusion of ≥ 2 units of packed read blood cells, or intracranial, intraspinal, intraocular, pericardial, retroperitoneal, intramuscular causing compartment syndrome, or fatal bleeding.
Clinical Relevant Non Major Bleeding (CRNMB) | From the date of index VTE to CRNMB occurrence, assessed up to 12 months
  CRNMB was defined as overt bleeding not meeting the criteria for MB but associated with medical intervention, unscheduled contact with a member of the health care team, temporary cessation of the treatment, or impairment of activities of daily life.

SECONDARY OUTCOMES:
All cause mortality | One year follow up since index VTE identified until the date of death from any cause, whichever came first, , assessed up to 12 months
  Deaths, regardless of the mechanism, were included in the all-cause mortality outcome

CONTACTS AND LOCATIONS:
Overall Officials: xiaoyan li, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No